CLINICAL TRIAL: NCT04407754
Title: Myo-Inositol as an Adjuvant to Letrozole for Infertility in PolyCystic Ovary Syndrome (MALI-PCOS): a Randomized Pilot Trial
Brief Title: Myo-Inositol for Infertility in PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12103
Record Dates: First submitted 2020-05-21; First posted 2020-05-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Placebo Comparator): This group will receive placebo powder twice daily.
  Interventions: Dietary Supplement: Placebo supplement
- Inositol Arm (Active Comparator): This group will receive myo-inositol (2,000mg) plus d-chiro-inositol (50mg) supplement powder twice daily.
  Interventions: Dietary Supplement: Inositol supplement

INTERVENTIONS:
Dietary Supplement: Inositol supplement — Inositol supplements given to inositol arm
  Arms: Inositol Arm
Dietary Supplement: Placebo supplement — Placebo supplement given to placebo arm
  Arms: Control Arm

SUMMARY:
This will be a prospective, double-blind randomized clinical trial of letrozole and placebo versus letrozole and inositols for up to 5 treatment cycles of ovulation induction or until pregnancy is achieved. All participants and members of the research team will be blinded to the treatment arms. Placebo and inositol supplement will be packaged to appear the same, tested, and packaged by a commercial supply company. The inositols will be a 40:1 blend of myo-inositol and D-chiro inositol.

DETAILED DESCRIPTION:
At the screening visit, blood pressure and heart rate will be measured, weight and height obtained and body mass index calculated (kg/m2). If not already completed at their new patient visit, transvaginal ultrasound will be performed to assess uterine anatomy and obtain antral follicle count, TSH, prolactin, and testosterone will be drawn, and serum samples will be obtained and analyzed for metabolic parameters (fasting lipids, insulin, and complete metabolic panel). One additional tube of blood will be drawn to store for potential future analysis. Once enrolled, randomization will occur and subjects will start either inositols or placebo. 84 women will be stratified by BMI and randomized 1:1 into two treatment arms, A) "Control Arm" = twice daily placebo powder and B) "Inositol Arm" = twice daily myo-inositol (2,000mg) plus d-chiro-inositol (50mg) supplement powder.

Treatment with either placebo or inositol will begin upon randomization. Participants will complete a validated quality of life in PCOS questionnaire (PCOSQ) at this visit and again upon study completion (11). Treatment with letrozole will begin after the baseline visit, which will occur after spontaneous menses or withdrawal bleeding induced by progestin administration. Because of this timing, participants will undergo pretreatment with inositol or placebo for a variable amount of time up to 6 weeks, with an anticipated average of 2-3 weeks. Metabolic parameters will be repeated after approximately 6 (7-9) and approximately 12 (11-13) weeks of inositol or placebo, at whichever study visit is most proximal in time to this goal timeframe. Both groups will receive letrozole 5mg every day for 5 days on days 3-7 of their menstrual cycle and instructed on timing intercourse with anticipated ovulation dates. Blood will be drawn for a serum progesterone each cycle between cycle days 20-22 to confirm ovulation, and repeated 1 week later if the initial progesterone level is below the threshold to confirm ovulation. Once ovulation is confirmed, they patient will expect a period 7-10 days later. They will call with cycle day 1 of bleeding if it occurs to start their next cycle of treatment, up to 5 cycles. If no bleeding occurs within the expected timeframe, they will check a home pregnancy test and call with results. Patients will complete medication side effect questionnaires at the first blood draw for progesterone of each cycle. This will be reviewed same-day and in person with the research nurse coordinator. Each patient will complete up to 5 cycles. Dose of letrozole will be increased in subsequent cycles for non-response or late ovulatory response (ovulation later than the progesterone blood draw) up to 10mg of letrozole a day. For patients with a second progesterone level below the threshold to confirm ovulation (day 21 and day 28), the higher dose of letrozole will be initiated following the receipt of the second low progesterone result. For patients who do not ovulate on the maximum dose of letrozole, their study participation will be considered complete.

Data to be collected will include: demographic information and medical history [age, race/ethnicity, body mass index (BMI), antral follicle count, length of infertility, prior infertility treatment (yes or no), obstetrical history, medical history, surgical history, current medication and allergy lists], partner information [age, race/ethnicity, BMI, general medical health assessment, prior paternity history], transvaginal ultrasound results, and serum studies [TSH, prolactin, progesterone, hCG levels, androgen levels (total and free testosterone, SHBG), and metabolic factors (fasting lipid panel, fasting glucose, fasting insulin, glucose:insulin ratio, HOMA-IR index)]. Questionnaires to be completed include: PCOSQ validated questionnaire for PCOS-related quality of life, and a side effect questionnaire about known side effects of letrozole and inositols. In addition to the baseline transvaginal ultrasound, additional ultrasounds may be performed as indicated clinically (including for establishing clinical pregnancy). Pertinent demographic and clinical information on patients who are participating in the study will be entered into a study database REDCap secure software.

Using the reported clinical pregnancy rate for infertile PCOS patients treated with letrozole of 31.3% (12) as the control group proportion (0.31) with a goal of 10% effect size (and therefore treatment group proportion 0.41), an alpha of 0.05, and power of 0.8, our sample size is estimated (for a full clinical trial) at ~361 in each arm. In considering the previously observed drop-out rate of ~20% in a similar patient population (3), we estimate that for a full clinical trial, we would need 452 participants randomized in each arm. Based on previously published literature regarding estimation of pilot randomized trial sample sizes, we will target 9% of this sample size for our pilot study to suggest or identify a significant difference (13). In conclusion, our planned study size will be 42 participants in each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Female patient age 18-36
* Desire for pregnancy
* Diagnosis of oligo- or anovulation secondary to polycystic ovary syndrome -All subjects must have ovulatory dysfunction and at least one of the remaining two criteria:hyperandrogenism or polycystic ovarian morphology on ultrasound
* At least one patent fallopian tube
* Normal uterine cavity
* Male partner with sperm concentration of at least 14 million/mL in at least one ejaculate.

Exclusion Criteria:

* Cause of anovulation other than PCOS such as uncontrolled thyroid dysfunction or hyperprolactinemia
* Presence of another major infertility factor
* Diabetes
* Contraindication to pregnancy
* Myo-inositol use < 3 months prior to study enrollment
* Concomitant metformin use. Previous use is allowed with last use at least 6 weeks prior to randomization.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | Through study completion, an average of 6 months
  Clinical pregnancy will be defined as documentation of a viable intrauterine pregnancy as noted by visualization of fetal heart motion on ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Burks, MD, Principal Investigator — OUHSC
Locations (1):
- OUHSC Reproductive Medicine Clinic, Oklahoma City, Oklahoma, United States